CLINICAL TRIAL: NCT03649568
Title: Effect of Consuming Ounce Equivalent Portions of Fresh Pork Versus Nuts, Beans, and Eggs as Defined by the Dietary Guidelines for Americans on Essential Amino Acid Substrate Availability for Protein Anabolism
Brief Title: Protein Source on Plasma Amino Acid Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1804020520
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Protein Deposition
MeSH Terms: interventions — Pork Meat; Eggs

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pork (Experimental): 1 ounce lean pork
  Interventions: Other: Pork
- Egg (Active Comparator): 1 large whole egg
  Interventions: Other: Egg
- Black beans (Experimental): 0.5 cups cooked black beans
  Interventions: Other: Black beans
- Almonds (Experimental): 1 ounce almonds
  Interventions: Other: Almonds

INTERVENTIONS:
Other: Pork — 1 oz lean pork
  Arms: Pork
Other: Egg — 1 large whole egg
  Arms: Egg
Other: Black beans — 0.5 cups cooked black beans
  Arms: Black beans
Other: Almonds — 1 oz almonds
  Arms: Almonds

SUMMARY:
This study will determine the effect of the same ounce-equivalents of fresh pork versus nuts, beans, and eggs on postprandial plasma essential amino acid availability in adults. Each participant will receive all four treatments.

DETAILED DESCRIPTION:
The 2015-2020 Dietary Guidelines for Americans stipulates how much Protein Foods should be consumed per day and per week as part of a Healthy U.S.-Style Eating Pattern. The predominant protein sources include lean meats, poultry, and eggs, however, nuts, seeds, and soy products are also included. Ounce-equivalents (oz-eq) are used as a standard unit of measure to compare animal to non-animal protein sources. One oz-eq of lean meat (1 oz) is equal to 0.5 oz of nuts (1 oz-eq), 0.25 cups (1 oz-eq) of beans, and one whole egg (1 oz-eq). One limitation of this unit of measure is that the protein quantity and quality of the foods are not considered. For example, 1 oz-eq of pork loin contains ~7 g of dietary protein whereas 1 oz-eq of almonds contains 3 g of protein. Consequently, consuming an oz-eq portion of protein foods from different sources could have different effects on the anabolic response to feeding. The purpose of this study is to assess the effect of consuming ounce equivalent portions of fresh pork versus nuts, beans, and eggs on essential amino acid substrate availability for protein anabolism. While it would seem intuitive that this research would show that higher protein intakes from pork and egg will lead to higher plasma essential amino acid responses, this research is paramount to addressing the shortcoming of using oz-eq to achieve the Dietary Guidelines for Americans recommendations for Protein Foods. This research will serve as an important resource for future Dietary Guidelines Advisory Committees to reevaluate the appropriateness of equating animal- and plant-based Protein Foods on the current ounce-equivalent basis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 25-39
* BMI 25-35 kg∙m-2
* Weight stable (± 4.5 kg) 3 months pre-study
* Not acutely ill
* Not diabetic
* Not pregnant or lactating
* Not currently (or within 3 months pre-study) following a vigorous exercise regimen
* Non-smoking
* Willing to consume study foods and travel to testing facilities.

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid concentrations | 5 hours
  Plasma samples will be drawn at times 0, 30, 60, 120, 180, 240, and 300 minutes after the consumption of the trial meal.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided